CLINICAL TRIAL: NCT03064399
Title: Microfracture Technique for the Treatment of Articular Cartilage Lesions of the Talus With or Without Lateral Ligament Repairment
Brief Title: Microfracture Technique for Talar Articular Cartilage Lesions With or Without Lateral Ligament Repairment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Responsible Party: Principal Investigator, Liming Cheng, Professor, Shanghai Tongji Hospital, Tongji University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 56014768-5
Record Dates: First submitted 2017-02-22; First posted 2017-02-27 (Actual); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Lateral Ligament Repair; Talar Cartilage Lesion; Microfracture
MeSH Terms: conditions — Fractures, Stress

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lateral ligament repairment (Experimental)
  Interventions: Procedure: lateral ligament repairment
- without lateral ligament repairment (Experimental)
  Interventions: Procedure: without lateral ligament repairment

INTERVENTIONS:
Procedure: without lateral ligament repairment — microfracture without repairment of the lateral ligament
  Arms: without lateral ligament repairment
Procedure: lateral ligament repairment — microfracture combined with repairment of the lateral ligament
  Arms: lateral ligament repairment

SUMMARY:
To study the clinical efficacy of microfracture combined with lateral ligament repairment for cartilage lesions of talus through the comparison between microfracture with and without lateral ligament repairment.

ELIGIBILITY:
Inclusion Criteria:

Full - thickness cartilage injury

Exclusion Criteria:

Age: > 40 years old or < 18 years old; BMI > 30; lesion > 4 cm2

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-02-28 (Estimated); Primary Completion 2019-05-28 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
Function score | One year after surgery
  AOFAS ankle function score

SECONDARY OUTCOMES:
Imaging result | One year after surgery
  Anatomical data from imaging results when bearing